CLINICAL TRIAL: NCT04222166
Title: Registry of Amniotic Membrane: Evaluating Utilization and Outcomes in Various Applications
Status: Completed | Type: Observational
Sponsor: MED Institute Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 19-003
Record Dates: First submitted 2020-01-03; First posted 2020-01-09 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Orthopedic Disorder; Wound
MeSH Terms: conditions — Musculoskeletal Diseases; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: CAM — Cryopreserved Amniotic Membrane

SUMMARY:
This registry will assess clinical outcomes following the use of Cryopreserved Amniotic Membrane (CAM) for the treatment of orthopedic and various other conditions. This registry will collect outcomes data via a registry of up to 100 patients who have received treatment with CAM in the post-market setting. Patients will be enrolled from up to five healthcare centers.

DETAILED DESCRIPTION:
The objective of this registry is to collect outcomes data via a registry on the uses of CAM in the post-market setting, including:

* Adverse events related to the treatment, or the product, will be collected for up to 12 weeks following the treatment.
* Improvements in appropriate effectiveness markers for CAM use in patients treated for various conditions.
* Improvements in overall quality of life resulting from CAM treatment in patients.

An additional objective is to determine standard of care follow-up for the target treatments, including effectiveness metrics used and typical follow-up schedule.

This registry is intended to collect clinical data from patients for analysis purposes only and will not be used to treat patients. The plan does not allow for any deviation from standard of care practice. Therefore, there is no added risk to patients from participating in the registry.

The sponsor will use an electronic data capture (EDC) system for capturing all the data from the sites. The system will be built and validated prior to initiation of the sites. Each participating physician or appropriately trained designee shall enter data into the EDC system, providing all applicable data and documentation to the sponsor. Data will be reviewed for missing data, data consistency, and reasonableness of responses. Discrepancies will be resolved through a formal query process within the EDC system, and may involve direct contact with hospital staff.

The conduct of the registry will be supervised through a process of centralized and on-site monitoring. The sponsor may remotely monitor the registry for data completeness and for adverse events. On-site monitoring will be implemented as necessary throughout the course of the registry. The physician/clinic will provide direct access to source data/documents for registry-related monitoring, audits and IRB review.

ELIGIBILITY:
Inclusion Criteria:

• A patient is suitable for inclusion in this registry if the patient has been treated with CAM for any indication as per the standard of care practice.

Exclusion Criteria:

• Patients are excluded from registry enrollment if they are under the age of 22 years.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A patient is suitable for inclusion in this registry if the patient has been treated with CAM for any indication as per the standard of care practice.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-08-06 (Actual)

PRIMARY OUTCOMES:
Incidence of related serious adverse events | 12 weeks
  Number of related serious adverse events occurred

SECONDARY OUTCOMES:
Visual Analog Scale | 12 weeks
  Change in pain score (0-10; higher scores mean worse outcome)
Change in analgesic use | 12 weeks
  Change in analgesic use
Change in wound size | 12 weeks
  Change in wound size
Time to complete wound closure | 12 weeks
  Time to complete wound closure

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Heise, PhD, Study Chair — MED Institute Inc.
Locations (2):
- United States (2):
  - Regenerative Medicine and Pain Management Physicians, Gulf Breeze, Florida
  - Foot and Ankle Specialists of South Jersey, Voorhees Township, New Jersey

IPD SHARING:
Plan to Share IPD: No